CLINICAL TRIAL: NCT02387983
Title: Pharmacokinetics and Safety of Solid Oral Posaconazole (MK-5592, POS) in Chinese Subjects at High Risk for Invasive Fungal Infections
Brief Title: Pharmacokinetics and Safety of Oral Posaconazole (MK-5592)Tablets in Chinese Participants at High Risk for Invasive Fungal Infections (MK-5592-117)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5592-117
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posaconazole (Experimental): Posaconazole 300 mg tablet (3 x 100 mg tablets) once every 12 hours on Day 1 and once-daily on Days 2 to 28
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — Posaconazole 300 mg solid oral tablet
  Other Names: MK-5592

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of oral posaconazole tablets in Chinese participants at high risk for invasive fungal infections. Neutropenic participants undergoing chemotherapy for acute myelogenous leukemia or myelodysplastic syndromes will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participant
* Female of reproductive potential with a serum hCG level consistent with a nongravid state and agree to use 2 acceptable methods of birth control throughout the study
* Body Mass Index (BMI) >=15 and <=30 kg/m^2
* Anticipated or documented prolonged neutropenia and likely to last for at least 7 days due to: a) standard intensive chemotherapy, anthracycline-based or other accepted regimen (excluding any investigational agent) for a new diagnosis of acute myelogenous leukemia (AML); b)chemotherapy for AML in first relapse; or c) therapy for myelodysplastic syndromes in transformation to AML or other diagnoses of secondary AML (therapy related, antecedent hematological disorders) or chronic myelogenous leukemia in blast crisis
* Free from any clinically significant disease other than the primary hematologic disease that would interfere with administration of study medication or study evaluations

Exclusion Criteria:

* Pregnant, intends to become pregnant during the study, or has been nursing
* Mentally or legally incapacitated, has significant emotional problems, or has clinically significant psychiatric disorder over the last 5 years
* Received systemic antifungal therapy (oral, intravenous, or inhaled) within 30 days of study enrollment for reasons other than antifungal prophylaxis
* Known or suspected invasive or systemic fungal infection
* Taken posaconazole within 10 days prior to study enrollment
* Major surgery, donated or lost 1 unit of blood, or participated in another investigational study within 4 weeks prior to the study
* Type 1 hypersensitivity or idiosyncratic reactions to azole agents
* Significant multiple or severe allergies, or has had an anaphylactic reaction or significant intolerability to drugs or food
* Moderate or severe liver dysfunction
* Chronic active hepatitis, cirrhosis, Hepatocellular Carcinoma (HCC), or other hepatic disease caused by a virus
* Previous electrocardiogram with a prolonged QTc interval
* Prior enrollment in this study or other posaconazole studies within 90 days of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status was >2 prior to induction chemotherapy for the underlying disease
* Known or suspected Gilbert's disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Liu K, Wu D, Li J, Chen H, Ning H, Zhao T, Dai H, Chen L, Mangin E, Winchell GA, Waskin H, Jiang J, Qiu Y, Zhao XM. Pharmacokinetics and Safety of Posaconazole Tablet Formulation in Chinese Participants at High Risk for Invasive Fungal Infection. Adv Ther. 2020 May;37(5):2493-2506. doi: 10.1007/s12325-020-01341-x. Epub 2020 Apr 22. PMID 32319040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult (18 to 70 years of age) male and female participants with neutropenia undergoing chemotherapy for acute myelogenous leukemia (AML) or myelodysplastic syndromes (MDS) were recruited at 4 sites in China.
Groups:
- Posaconazole: All participants received posaconazole 300 mg tablet (3 x 100 mg tablets) once every 12 hours on Day 1 and once-daily on Days 2 to 28. The first 20 participants (Intensive and Sparse PK subgroup) underwent intensive and sparse pharmacokinetic (PK) sampling on Days 1 and 8; the next 45 participants (Sparse PK subgroup) underwent PK sampling on Day 8 only.
Period: Overall Study
Arm/Group | Posaconazole
Started | 65
Completed | 58
Not Completed | 7
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Posaconazole
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Average Concentration (ssCavg) of Posaconazole on Day 8
Description: The ssCavg was calculated in order to determine the percentage of participants achieving the pharmacokinetic (PK) target of ssCavg >500 ng/mL on Day 8 when plasma drug levels had reached steady state.
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 8
Population: The PK analysis set included all randomized and treated participants who complied with the protocol and have documented adherence to daily dosing and PK regimens through the Day 8 steady-state evaluation and have data available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 44
Percentage of Participants
  ssCavg < 500 ng/mL | 0.0
  500 ng/mL ≤ ssCavg < 2500 ng/mL | 88.9
  2500 ng/mL ≤ ssCavg < 3750 ng/mL | 11.1
  ssCavg ≥ 3750 ng/mL | 0

2. Primary Outcome: Steady-state Area Under the Concentration-time Curve (ssAUC0-24hr) of Posaconazole on Day 8
Description: The ssAUC0-24hr was calculated to determine the mean plasma drug concentration in the Intensive and Sparse PK subgroup from immediately after dosing to 24 hours post-dose on Day 8. Results data are presented as the arithmetic mean (% arithmetic coefficient of variation [CV]), where CV is calculated as (100 x standard deviation/arithmetic mean).
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 8
Population: The PK analysis set included all randomized and treated participants in the Intensive and Sparse PK subgroup who complied with the protocol and have documented adherence to daily dosing and PK regimens through the Day 8 steady-state evaluation and have data available.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 18
hr*ng/mL | 38600 (42.8)

3. Primary Outcome: Steady-state Maximum Concentration (ssCmax) of Posaconazole on Day 8
Description: The ssCmax was calculated in order to determine the maximum post-dose plasma drug concentration in the Intensive and Sparse PK subgroup on Day 8. Results data are presented as the arithmetic mean (% arithmetic coefficient of variation [CV]), where CV is calculated as (100 x standard deviation/arithmetic mean).
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 8
Population: The PK analysis set included all randomized and treated participants in the Intensive and Sparse PK subgroup who complied with the protocol and have documented adherence to daily dosing and PK regimens through the Day 8 steady-state evaluation with available data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 18
ng/mL | 2150 (43.9)

4. Primary Outcome: Steady-state Minimum Concentration (ssCmin) of Posaconazole on Day 8
Description: The ssCmin was calculated in order to determine the lowest measurable drug concentration in the Intensive and Sparse PK subgroup up to 24 hours post-dose on Day 8. Results data are presented as the arithmetic mean (% arithmetic coefficient of variation [CV]), where CV is calculated as (100 x standard deviation/arithmetic mean).
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 8
Population: The PK analysis set included all randomized and treated participants in the Intensive and Sparse subgroup who complied with the protocol and have documented adherence to daily dosing and PK regimens through the Day 8 steady-state evaluation with available data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 18
ng/mL | 1310 (43.6)

5. Primary Outcome: Time to Steady-state Maximum Concentration (ssTmax) of Posaconazole on Day 8
Description: The ssTmax was calculated in order to determine the amount of time required to reach ssCmax in the Intensive and Sparse PK subgroup on Day 8.
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 8
Population: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | Posaconazole
Number analyzed (Participants) | 18
hr | 4.04 [0.00 to 8.00]

6. Primary Outcome: AUC0-24hr of Posaconazole on Day 1
Description: The AUC0-24hr was calculated to determine the mean plasma drug concentration from immediately after dosing to 24 hours post-dose in the Immediate and Sparse PK subgroup on Day 1. Results data are presented as the arithmetic mean (% arithmetic coefficient of variation [CV]), where CV is calculated as (100 x standard deviation/arithmetic mean).
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 20
hr*ng/mL | 14500 (39.0)

7. Primary Outcome: Cmax of Posaconazole on Day 1
Description: The Cmax was calculated to determine the maximum plasma drug concentration up to 24 hours post-dose in the Immediate and Sparse PK subgroup on Day 1. Results data are presented as the arithmetic mean (% arithmetic coefficient of variation [CV]), where CV is calculated as (100 x standard deviation/arithmetic mean).
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1
Population: The PK analysis set included all randomized and treated participants in the Immediate and Sparse PK subgroup who complied with the protocol and have documented adherence to daily dosing and PK regimens through the Day 8 steady-state evaluation with available data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 20
ng/mL | 730 (47.7)

8. Primary Outcome: Cmin of Posaconazole on Day 1
Description: The Cmin was calculated in order to determine the lowest measurable drug concentration from immediately after dosing to 24 hours post-dose in the Immediate and Sparse PK subgroup on Day 1. Results data are presented as the arithmetic mean (% arithmetic coefficient of variation [CV]), where CV is calculated as (100 x standard deviation/arithmetic mean).
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 20
ng/mL | 997 (35.9)

9. Primary Outcome: Tmax of Posaconazole on Day 1
Description: The Tmax was calculated in order to determine the time required to reach Cmax in the Immediate and Sparse PK subgroup on Day 1.
Time Frame: Pre-dose and 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Posaconazole
Number analyzed (Participants) | 20
Hours | 3.99 [1.97 to 7.98]

ADVERSE EVENTS:
Time Frame: Up to Day 42
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Groups:
- MK-5592: All participants received posaconazole 300 mg tablet (3 x 100 mg tablets) once every 12 hours on Day 1 and once-daily on Days 2 to 28. The first 20 participants (Intensive and Sparse group) underwent intensive and sparse PK sampling on Days 1 and 8; the next 45 participants (Sparse group) underwent PK sampling on Day 8 only.
Arm/Group | MK-5592
Serious Adverse Events (participants affected / at risk) | 4/65
Other Adverse Events (participants affected / at risk) | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5592 (N=65)
Anal infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5592 (N=65)
Anaemia (Blood and lymphatic system disorders) | 6 (16)
Leukopenia (Blood and lymphatic system disorders) | 11 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (32)
Abdominal discomfort (Gastrointestinal disorders) | 4 (5)
Abdominal distension (Gastrointestinal disorders) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 22 (25)
Faeces hard (Gastrointestinal disorders) | 4 (4)
Mouth ulceration (Gastrointestinal disorders) | 7 (10)
Nausea (Gastrointestinal disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 4 (4)
Asthenia (General disorders) | 6 (7)
Chest discomfort (General disorders) | 5 (5)
Oedema peripheral (General disorders) | 10 (13)
Pyrexia (General disorders) | 35 (59)
Febrile infection (Infections and infestations) | 6 (8)
Lung infection (Infections and infestations) | 11 (12)
Soft tissue infection (Infections and infestations) | 5 (7)
Transfusion related complication (Injury, poisoning and procedural complications) | 5 (10)
Alanine aminotransferase increased (Investigations) | 12 (12)
Aspartate aminotransferase increased (Investigations) | 8 (8)
Blood bilirubin increased (Investigations) | 14 (17)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 15 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (32)
Hypoproteinaemia (Metabolism and nutrition disorders) | 10 (11)
Dizziness (Nervous system disorders) | 5 (6)
Insomnia (Psychiatric disorders) | 4 (5)
Haematuria (Renal and urinary disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 14 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.